CLINICAL TRIAL: NCT04723680
Title: An Exploration of the Impact of Gene Therapy on the Lives of People With Haemophilia and Their Families
Acronym: Exigency
Status: Completed | Type: Observational
Sponsor: Haemnet (Other)
Collaborators: UniQure Biopharma B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: v3Nov2020
Record Dates: First submitted 2021-01-15; First posted 2021-01-26 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hemophilia
Keywords: Haemophilia, Gene Therapy, Quality of Life
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Early dose finding cohort: People with Haemophilia who took part in the early dose finding studies
  Interventions: Other: Qualitative interview
- Subsequent studies group cohort: People with haemophilia who took part in subsequent gene therapy studies
  Interventions: Other: Qualitative interview
- Withdrawn/ineligible Cohort: People with haemophilia who were withdrawn or proved ineligible
  Interventions: Other: Qualitative interview
- Not interested cohort: People with haemophilia who are definitely not interested in gene therapy
  Interventions: Other: Qualitative interview
- Not offered cohort: People with haemophilia who are interested in gene therapy but have not been the opportunity to take part
  Interventions: Other: Qualitative interview

INTERVENTIONS:
Other: Qualitative interview — Qualitative semi structured interview

SUMMARY:
This study programme aims to examine the real-world experience and impact of gene therapy in a diverse community of people and families affected by haemophilia who have been or will be exposed to gene therapy.

DETAILED DESCRIPTION:
This is a prospective observational multiple cohort qualitative research study to be conducted among diverse groups within the haemophilia community whose lives may have been impacted by gene therapy.

The study is designed to allow English-speaking patients and their families to tell their own life stories through narrative accounts. The narratives represent a true sharing of experiences and offer insight into how these patients and families cope with haemophilia.

ELIGIBILITY:
Inclusion Criteria:

* People with haemophilia A or B who consented to and have undergone gene therapy in the early dose-finding studies and a member of their family
* People with haemophilia A or B who consented to a gene therapy trial following the results of the early studies and a member of their family
* People with haemophilia A or B who consented to a gene therapy trial but who withdrew, were withdrawn from, or were ineligible for the study, and a member of their family
* People with haemophilia A or B who are definitely not interested in or unaware of gene therapy and a member of their family
* People with haemophilia A or B who are interested in but have not been offered gene therapy
* Those who have given written consent to be in the study
* All participants will be ≥16 years.

Exclusion Criteria:

* Participants will be excluded if they do not speak English (for the interviews) or do not consent to be in the study.

Ages: 16 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with haemophilia and a member of their family
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
patient expectations | Each participant & family member will take part in a 1 hour semi structured qualitative interview where his experiences of his condition, previous treatment & experience of gene therapy will be discussed & analysed using a grounded theory approach
  To explore the expectations that patients, and families in the UK have of gene therapy and its position in contemporary and future haemophilia management

SECONDARY OUTCOMES:
Lived experience | Each participant & family member will take part in a 1 hour semi structured qualitative interview where his experiences of his condition, previous treatment & experience of gene therapy will be discussed & analysed using a grounded theory approach
  To understand the lived experience of people who have undergone gene therapy
Impact of gene therapy | Each participant & family member will take part in a 1 hour semi structured qualitative interview where his experiences of his condition, previous treatment & experience of gene therapy will be discussed & analysed using a grounded theory approach
  To understand the as yet "unseen" impact of gene therapy on the extended family
Impact of ineligibility | Each participant & family member will take part in a 1 hour semi structured qualitative interview where his experiences of his condition, previous treatment & experience of gene therapy will be discussed & analysed using a grounded theory approach
  To understand the impact of ineligibility for gene therapy trials
Impact of withdrawal | Each participant & family member will take part in a 1 hour semi structured qualitative interview where his experiences of his condition, previous treatment & experience of gene therapy will be discussed & analysed using a grounded theory approach
  To understand the impact of withdrawal from gene therapy on individuals and their ongoing attitude to their haemophilia care
Why not interested | Each participant & family member will take part in a 1 hour semi structured qualitative interview where his experiences of his condition, previous treatment & experience of gene therapy will be discussed & analysed using a grounded theory approach
  To understand why some patients and families opt not to participate in gene therapy trials as a treatment option

CONTACTS AND LOCATIONS:
Overall Officials: Simon P Fletcher, Principal Investigator — Researcher
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT04723680/Prot_000.pdf